CLINICAL TRIAL: NCT00979888
Title: A Non-pharmacological Supportive Care Intervention for Patients With Lung Cancer and Their Caregivers in the Management of the Respiratory Distress Symptom Cluster.
Brief Title: Study of How Caregivers Help Patients Cope With Respiratory and Other Symptoms Caused by Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000649867; UM-LC-Symptom-Clusters; EU-20972
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Anxiety Disorder; Depression; Dyspnea; Fatigue; Lung Cancer
Keywords: dyspnea; depression; fatigue; anxiety disorder; small cell lung cancer; non-small cell lung cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Dyspnea; Fatigue; Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Psychiatric Rehabilitation; Caregivers

INTERVENTIONS:
Other: educational intervention
Other: informational intervention
Other: psychosocial support for caregiver
Other: questionnaire administration
Procedure: dyspnea management
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Gathering information about how patients, caregivers, and healthcare professionals cope with symptoms caused by lung cancer, such as breathlessness, cough, fatigue, anxiety, depression, pain, and difficulty sleeping, may help doctors learn more about non-drug methods of treating symptoms of respiratory distress.

PURPOSE: This clinical trial is studying how caregivers help patients cope with respiratory and other symptoms caused by lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To consolidate knowledge of existing interventions and their characteristics.
* To seek patients', caregivers', and healthcare professionals' views on existing interventions and to establish whether these groups utilize any additional interventions not currently described in the literature.
* To explore patients' perspectives on interrelationships among symptoms, in terms of clusters or causal relationships.
* To identify patients', caregivers', and healthcare professionals' views of the desirable components/characteristics of a novel intervention.
* Explore what is 'usual care' in the context of the study.

OUTLINE: This is a multicenter study.

The management of cough and breathlessness in respiratory diseases and lung cancer is assessed through a narrative review of interventions to support caregivers in providing physical care to patients with cancer and explore qualitative patient symptom experience with a particular focus on identifying specific characteristics and components of interventions and identifying patients' and caregivers' explanations of how the respiratory symptom cluster relates to other symptom experiences (e.g., fatigue, depression, anxiety).

Patients and caregivers undergo 2-3 face-to-face interviews to assess views on existing interventions in terms of perceived effectiveness, acceptability, importance, and feasibility; to establish whether additional interventions (formal or self-initiated) are employed; to address patient and caregiver experiences of symptom interactions and clusters; and to fine tune the content of the planned intervention and identify any synergies between symptoms as discussed by patients. Healthcare professionals undergo similar assessments via focus groups.

Patient and caregiver views on desirable components of a novel intervention are assessed by means of Discrete Choice Experiment (DCE) using a 'Best-Worst Scaling' (BWS) approach to allow identification of the relative importance of several attributes by means of a series of scenarios to enable a focus on characteristics of a nonpharmacological intervention, rather than requiring respondents to make judgments about the usefulness of specific interventions (e.g., counseling, aromatherapy) with which they may be unfamiliar.

PROJECTED ACCRUAL: This study will accrue 30-40 pairs of patients and caregivers.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patient with diagnosis of lung cancer
  * Caregiver of patient
  * Healthcare professional (i.e., clinical nurse specialist, physiotherapist, primary care team member, or palliative care team member)
* Patients recruited from Manchester, Liverpool, or Southampton hospitals

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Consolidation of knowledge of existing interventions and their characteristics
Patients', caregivers', and healthcare professionals' views on existing interventions
Utilization of any additional interventions not currently described in the literature
Exploration of patients' perspectives on interrelationships among symptoms, in terms of clusters or causal relationships
Patients', caregivers', and healthcare professionals' views of the desirable components/characteristics of a novel intervention using the Discrete Choice Experiment 'Best-Worst' scale
Exploration of what is 'usual care' in the context of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, MD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, England, United Kingdom